CLINICAL TRIAL: NCT00714727
Title: Set Point Acupuncture for Migraines Using a Digital Assistant
Acronym: SPAMDA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC 07-12
Record Dates: First submitted 2008-07-10; First posted 2008-07-14 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2009-09

CONDITIONS: Migraine Headaches
Keywords: migraine; headache; acupuncture
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — 8 weeks of acupuncture, starting with twice a week for 4 weeks, followed by once a week for 4 weeks, using 8 standardized, bilateral acupuncture points.
  Other Names: Migraines

SUMMARY:
The object of this research study is to test a standardized set of acupuncture points on migraine patients to reduce frequency and intensity of headaches. Acupuncture has been studied in prior research but the treatment points have varied between subjects, making it difficult to replicate studies.

DETAILED DESCRIPTION:
Subjects will be recording daily headache activity on personal digital assistants (PDA's) for 12 weeks before and 12 weeks after 8 weeks of acupuncture intervention. MIDAS, HIT-6 and BDI-II measurements will be done at the beginning of the study (12 weeks pre-intervention), directly before the intervention, directly after, and 12 weeks post-intervention. Measurements will be compared before and after intervention. This is a follow-up to a successful earlier study when these same acupuncture points were used on subjects with chronic daily headache, the majority being migraine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 21 years and 65 years of age
* Subjects with a history of migraine headaches for at least 12 months
* Subjects who have not received acupuncture for any medical condition in the past 6 months.
* A negative pregnancy test for childbearing females since some acupuncture points may be contraindicated in pregnancy. Pregnancy tests will be conducted at MMC.
* Subjects willing and able to use a PDA daily for data collection

Exclusion Criteria:

* Subjects who plan to receive acupuncture treatment for any other type of medical condition while enrolled in this protocol
* Subjects with the presence of organic pathology (i.e., brain tumor)
* Subjects who have the presence of a systemic disorder or illness, including serious psychiatric illness
* Subjects who began a new headache treatment less than two weeks before proposed enrollment date
* Subjects who are pregnant, lactating, or planning to become pregnant within 6 months
* Subjects that use alcohol on a regular basis
* Subjects that use recreational drugs
* Subjects that have a cardiac pacemaker
* Subjects that use analgesics on more than 10 days per month
* Subjects that exercise prophylactic headache treatment with drugs during the past 4 weeks

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
If a standard set of acupuncture points delivered over a set time frame, reduces the frequency and intensity of headaches in a population of migraine sufferers. | 32 weeks

SECONDARY OUTCOMES:
Measurements of the impact of acupuncture intervention will be detected when baseline measurements of frequency and severity of headaches is compared to measurements taken 12 weeks after the last acupuncture session. MIDAS, HIT-6, BDI-II and SF-12 scores | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Plank, MD, LAc, Principal Investigator — John P. Murtha Neuroscience and Pain Institute
Locations (1):
- John P Murtha Neuroscience and Pain Institute, Johnstown, Pennsylvania, United States